CLINICAL TRIAL: NCT04668066
Title: A PHASE 1 FIRST IN HUMAN, RANDOMIZED, DOUBLE BLIND, SPONSOR OPEN, PLACEBO-CONTROLLED, SINGLE- AND MULTIPLE DOSE ESCALATION, PARALLEL GROUP STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF 07242813 IN HEALTHY PARTICIPANTS AND PARTICIPANTS WITH ATOPIC DERMATITIS
Brief Title: Study to Evaluate Safety and Tolerability of PF-07242813 in Healthy Participants and Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C4461001
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; inflammatory skin disease
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single ascending doses of PF-07242813 or placebo in healthy participants (Experimental): Participants will receive a single intravenous dose of either PF-07242813 or placebo
  Interventions: Drug: PF-07242813; Drug: Placebo
- Multiple ascending doses of PF-07242813 or placebo in healthy participants (Experimental): Participants will receive multiple subcutaneous doses PF-07242813 or placebo
  Interventions: Drug: PF-07242813; Drug: Placebo
- Single dose of PF-07242813 or placebo in participants with moderate to severe atopic dermatitis (Experimental): Participants will receive a single intravenous dose of either PF-07242813 or placebo
  Interventions: Drug: PF-07242813; Drug: Placebo

INTERVENTIONS:
Drug: PF-07242813 — PF-07242813 given intravenously or subcutaneous
Drug: Placebo — Placebo given intravenously or subcutaneous

SUMMARY:
This is the first time PF-07242813 will be given to humans. The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of escalating single and repeat doses of PF-07242813 in healthy participants and in participants with moderate to severe atopic dermatitis. An additional goal is to assess the pharmacodynamics of PF-07242813 in participants with moderate to severe AD, including potential effects on clinical signs and symptoms.

ELIGIBILITY:
Inclusion Criteria Part 1 (Healthy Volunteer Cohorts):

* BMI of 17.5 to 30.5 kg/m2; and BW>50 kg (110 lbs)
* Overtly healthy as determined by medical evaluation including medical history, physical examination, vital sign assessments, temperature, 12-lead ECGs, laboratory tests
* Japanese cohort: healthy adults of Japanese descent, where parents and grandparents are Japanese
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol

Inclusion Criteria Part 2 (Atopic Dermatitis Cohort):

* Have a clinical diagnosis of chronic atopic dermatitis (also known as atopic eczema) for approximately 1 year prior to Day 1 and have the diagnosis of AD confirmed (Hanifin and Rajka criteria of AD).
* Either have had an inadequate response to treatment with topical medications (for at least 4 consecutive weeks within 1 year of the first dose of the study drug) OR Have a documented reason why topical treatments are considered medically inappropriate (eg, because of important side effects or safety risks) within the last year.
* Have moderate to severe AD (defined as having an affected BSA (captured as part of EASI) ≥10%, IGA ≥3, and EASI ≥12 at both the screening and baseline visits).
* Generally healthy adult, with no significant comorbidities.
* Mild or moderate asthma that is well-controlled (not requiring high dose inhaled corticosteroids, systemic [oral or parenteral] corticosteroids, or biologic asthma treatments).
* BMI of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria Part 1 (Healthy Volunteer Cohorts):

* Evidence of active, latent, or inadequately treated infection with TB; History of HIV, hepatitis B or C infection; positive testing for HIV, HepB, HepC except HepB vaccination
* Medical or psychiatric condition that may increase the risk of study participation, or inappropriate for the study in investigator's judgement
* History of any lymphoproliferative disorder, evidence or history of clinically significant diseases
* History of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or judged clinically significant by the investigator within 6 months
* Known history of or evidence of current endocrine disease
* Exposure to live or attenuated vaccines within 28 days of screening.
* Have any malignancies or a history of malignancies except adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Have undergone significant trauma or major surgery within 1 month of 1st dose of study drug.
* Use of prescription or nonprescription drugs, dietary or herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to 1st dose of study drug.
* Females taking hormone replacement therapy may be eligible to participate in this study if they are willing to discontinue therapy at least 28 days prior to the first dose of study treatment and remain off hormonal therapy for the duration of the study.
* Positive urine drug test, alcohol intake more than 14 units per week or use of tobacco/nicotine containing products more than 5 cigarettes per day.
* Treatment with an investigational drug within 28 days or 5 half-lives preceding the first dose of study treatment (whichever is longer).
* Abnormal BP, ECG and lab tests including AST/ALT, total bilirubin and anterior pituitary hormones, at screenings and/or baseline, based on pre-specified criteria per protocol.
* Unwilling or unable to comply with the Lifestyle guidance specified in this protocol (Lifestyle Considerations section).

Exclusion Criteria Part 2 (Atopic Dermatitis Cohort):

* Evidence of active, latent, or inadequately treated TB.
* History of or positive result for HIV or hepatitis infection. Positive Covid-19 test (if collected).
* Significant medical or psychiatric condition, including suicidal ideation (C-SSRS screening assessment noting suicidal ideation in prior 6 months is not eligible).
* H/o or current endocrine disease.
* History of systemic infection requiring hospitalization, parenteral antimicrobial treatment or considered significant by Investigator.
* History of or current malignancy, with the exception of non-metastatic BCC, squamous cell skin or cervical in situ.
* Currently have active forms of other inflammatory skin diseases.
* Have history of or current evidence of skin disease at the time of Day 1 that would interfere with evaluation of atopic dermatitis or response to treatment.
* Have active chronic or acute skin infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to Day 1, or superficial skin infections within 1 week prior to Day 1.
* Score of >5 on the Fitzpatrick Skin Type Assessment.
* History of anaphylaxis with the exception of participants with sensitivity and/or anaphylaxis only to a single, avoidable allergen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - First OC Dermatology, Fountain Valley, California
  - Keck School of Medicine of USC, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Aspen Clinical Research, Orem, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4461001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts: Part 1 was conducted in healthy adult participants and Part 2 was conducted in adult participants with moderate to severe atopic dermatitis (AD).
Pre-assignment Details: A total of 122 participants (57 participants in single ascending dose [SAD] cohorts, 40 in multiple ascending dose [MAD] cohorts and 25 in AD cohorts) were enrolled across 5 centers in the United States.
Groups:
- Part 1: 0.3 mg IV SAD: Healthy participants were administered a single dose of 0.3 milligrams (mg) PF-07242813 as an intravenous (IV) infusion.
- Part 1: 1mg IV SAD: Healthy participants were administered a single dose of 1 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 3 mg IV SAD: Healthy participants were administered a single dose of 3 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 10 mg IV SAD: Healthy participants were administered a single dose of 10 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 30 mg IV SAD: Healthy participants were administered a single dose of 30 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 100 mg IV SAD: Healthy participants were administered a single dose of 100 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 300 mg IV SAD: Healthy participants were administered a single dose of 300 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 1000 mg IV SAD: Healthy participants were administered a single dose of 1000 mg PF-07242813 as an intravenous (IV) infusion.
- Part 1: 1000 mg IV SAD (Japanese Cohort): Healthy Japanese participants were administered a single dose of 1000 mg PF-07242813 as an IV infusion.
- Part 1: 15 mg SC Q2W MAD: Healthy participants were administered 15 mg PF-07242813 subcutaneously every 2 weeks (Q2W) for a total of 3 doses.
- Part 1: 50 mg SC Q2W MAD: Healthy participants were administered 50 mg PF-07242813 subcutaneously every 2 weeks (Q2W) for a total of 3 doses.
- Part 1: 150 mg SC Q2W MAD: Healthy participants were administered 150 mg PF-07242813 subcutaneously every 2 weeks (Q2W) for a total of 3 doses.
- Part 1: 300 mg SC Q2W MAD: Healthy participants were administered 300 mg PF-07242813 subcutaneously every 2 weeks (Q2W) for a total of 3 doses.
- Part 1: 500 mg IV Q2W MAD: Healthy participants were administered 500 mg PF-07242813 as IV infusion every 2 weeks (Q2W) for a total of 3 doses.
- Part 1: Placebo SAD: Healthy participants were administered a single dose of placebo as an IV infusion.
- Part 1: Placebo SC MAD: Healthy participants were administered placebo every 2 weeks (Q2W) for a total of 3 doses via the SC route.
- Part 1: Placebo IV MAD: Healthy participants were administered placebo every 2 weeks (Q2W) for a total of 3 doses as an IV infusion.
- Part 2: 1000 mg IV AD: Participants with atopic dermatitis were administered a single dose of 1000 mg PF-07242813 administered as an IV Infusion.
- Part 2: Placebo IV AD: Participants with atopic dermatitis were administered a single dose of placebo as an IV infusion.
Period: Part 1: Treatment Phase
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Started | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 17 | 8 | 2 | 0 | 0
Completed | 2 | 2 | 1 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 4 | 4 | 6 | 17 | 6 | 2 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part 1: Follow-Up
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Started | 2 | 2 | 1 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 (Eligible participants entered follow-up following discontinuation of study treatment.) | 6 (Eligible participants entered follow-up following discontinuation of study treatment.) | 6 | 17 | 8 (Eligible participants entered follow-up following discontinuation of study treatment.) | 2 | 0 | 0
Completed | 2 | 2 | 1 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 4 | 4 | 6 | 17 | 6 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part 2: Treatment Phase
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 (Participants enrolled in Part 2 of the study.) | 9 (Participants enrolled in Part 2 of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2: Follow-Up
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 8 (Eligible participants entered follow-up following discontinuation of study treatment.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants randomly assigned to study intervention and who received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 17 | 8 | 2 | 16 | 9 | 122
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 Years | 2 | 2 | 2 | 5 | 4 | 4 | 4 | 3 | 3 | 2 | 3 | 5 | 6 | 2 | 8 | 5 | 1 | 14 | 9 | 84
  45 to 64 Years | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 1 | 4 | 3 | 1 | 0 | 4 | 9 | 3 | 1 | 2 | 0 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 4 | 2 | 0 | 4 | 4 | 28
  Male | 1 | 2 | 2 | 6 | 5 | 3 | 4 | 5 | 2 | 6 | 5 | 4 | 6 | 5 | 13 | 6 | 2 | 12 | 5 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 2 | 0 | 1 | 3 | 1 | 2 | 1 | 6 | 1 | 1 | 3 | 2 | 36
  Not Hispanic or Latino | 1 | 1 | 0 | 4 | 4 | 4 | 3 | 4 | 4 | 5 | 3 | 5 | 4 | 5 | 11 | 7 | 1 | 13 | 7 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 2 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 2 | 0 | 3 | 3 | 3 | 4 | 0 | 1 | 6 | 2 | 31
  White | 2 | 2 | 2 | 5 | 2 | 4 | 3 | 4 | 0 | 4 | 6 | 2 | 3 | 2 | 10 | 7 | 1 | 6 | 4 | 69
  More than one race | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: SAD Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or other important medical events. An AE was considered as treatment emergent if the event started during the effective duration of treatment. All events that started on or after the first dosing day up to the last dose plus the lag time were considered as TEAEs.
Time Frame: From start of study treatment on Day 1 to Day 71
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: Placebo SAD
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 17
Participants
  TEAEs | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 2 | 6
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Part 1: MAD Cohorts: Number of Participants With TEAEs and TESAEs
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or other important medical events. An AE was considered as treatment emergent if the event started during the effective duration of treatment. All events that started on or after the first dosing day up to the last dose plus the lag time were considered as TEAEs.
Time Frame: From start of study treatment on Day 1 to Day 99
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
Participants
  TEAEs | 3 | 1 | 4 | 2 | 2 | 5 | 1
  TESAEs | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Part 2: Number of Participants With TEAEs and TESAEs
Description: as for outcome 2
Time Frame: From start of study treatment on Day 1 to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Number analyzed (Participants) | 16 | 9
Participants
  TEAEs | 4 | 5
  TESAEs | 0 | 1

4. Primary Outcome: Part 1: SAD Cohorts: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Vital signs included blood pressure, pulse rate, respiratory rate and temperature. Temperature was measured by oral, tympanic, or temporal artery method. Blood pressure and respiratory rate were measured with the participant in a supine position after 5 minutes of rest for the participant. Clinically significant findings were determined by the investigator.
Time Frame: From initiation of treatment to day 71
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: Placebo SAD
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 1: MAD Cohorts: Number of Participants With Clinically Significant Findings in Vital Signs
Description: as for outcome 4
Time Frame: From start of study treatment on Day 1 to Day 99
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part 2: Number of Participants With Clinically Significant Findings in Vital Signs
Description: as for outcome 4
Time Frame: From start of study treatment on Day 1 to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Number analyzed (Participants) | 16 | 9
Participants | 0 | 0

7. Primary Outcome: Part 1: SAD Cohorts: Number of Participants With Laboratory Test Abnormalities
Description: Pre-defined criteria for laboratory parameters were hemoglobin (HGB) (<0.8* Lower limit normal (LLN)), Erythrocyte (Ery). Mean Corpuscular (MC) Volume (<0.9* LLN), Ery MC Hemoglobin (<0.9* LLN), Ery. MC HGB Concentration (<0.9* LLN), Leukocytes (<0.6* LLN), Neutrophils (<0.8* LLN), Bilirubin (>1.5* Upper limit normal (ULN)), Aspartate Aminotransferase (>3.0* ULN), Urea Nitrogen (>1.3* ULN), Creatinine (>1.3* ULN), Urate (>1.2* ULN). Number of participants with any laboratory test abnormalities meeting pre-defined criteria was reported in this outcome measure.
Time Frame: Baseline (last pre-dose measurement) to Day 71
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: Placebo SAD
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 17
Participants | 1 | 1 | 1 | 2 | 2 | 3 | 3 | 4 | 2 | 12

8. Primary Outcome: Part 1: MAD Cohorts: Number of Participants With Laboratory Test Abnormalities
Description: Pre-defined criteria for laboratory parameters were HGB (<0.8* LLN), Ery MCV (<0.9* LLN), Ery MC Hemoglobin (<0.9* LLN), Ery. MC HGB Concentration (<0.9* LLN), Leukocytes (<0.6* LLN), Neutrophils (<0.8* LLN), Bilirubin (>1.5* ULN), Aspartate Aminotransferase (>3.0* ULN), Urea Nitrogen (>1.3* ULN), Creatinine (>1.3* ULN), Urate (>1.2* ULN). Number of participants with any laboratory test abnormalities meeting pre-defined criteria was reported in this outcome measure.
Time Frame: Baseline (last pre-dose measurement) to Day 99
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
Participants | 3 | 2 | 5 | 5 | 4 | 6 | 2

9. Primary Outcome: Part 2: Number of Participants With Laboratory Test Abnormalities
Description: as for outcome 8
Time Frame: Baseline (last pre-dose measurement) to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Number analyzed (Participants) | 16 | 9
Participants | 11 | 9

10. Primary Outcome: Part 1: SAD Cohorts Only: Number of Participants With Cardiac Telemetry Abnormalities
Description: Cardiac telemetry was collected in Part 1 SAD cohorts only. Number of participants with any cardiac telemetry abnormalities were reported in this outcome measure.
Time Frame: From pre-dose up to 6 hours post dose on Day 1
Population: Safety analysis set consisted of all participants randomly assigned to study intervention and who received at least one dose of study intervention. This outcome was planned to be analyzed for SAD cohorts only as pre-specified in protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: Placebo SAD
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Part 1: SAD Cohorts: Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG)
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, corrected QT (QTc) intervals and QRS complex. ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position. Clinically significant findings were determined by the investigator.
Time Frame: From pre-dose on Day 1 up to Day 71
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: Placebo SAD
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 1: MAD Cohorts: Number of Participants With Clinically Significant Findings in ECG
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, QTc intervals and QRS complex. ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position. Clinically significant findings were determined by the investigator.
Time Frame: From pre-dose on Day 1 up to Day 99
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part 2: Number of Participants With Clinically Significant Findings in ECG
Description: as for outcome 12
Time Frame: From pre-dose on week 1 to week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Number analyzed (Participants) | 16 | 9
Participants | 0 | 0

14. Secondary Outcome: Part 1: SAD Cohorts: Area Under the Serum Concentration Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) for PF-07242813
Description: AUClast was calculated using the linear/log trapezoidal method.
Time Frame: Pre-dose, 2, 6, 12, 24, 48, 72, 96, 336, 672 hours post-dose (for all cohorts); 1008 hours post-dose for all cohorts except 0.3 mg IV; 1344 and 1680 hours post-dose for all cohorts except 0.3 mg IV and 1 mg IV
Population: The PK parameter set consisted of all randomized participants who received at least 1 dose of study intervention and who have at least 1 of the PK parameters of interest calculated. Data was not summarized for PK parameters if less than 3 participants had evaluable data values as pre-specified in the statistical analysis plan; hence, individual values were reported for 0.3 mg IV SAD, 1 mg IV SAD and 3 mg IV SAD cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort)
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4
Nanogram*hour/milliliter | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 2390 and 3710. | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 14700 and 17500. | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 55100 and 80800. | 546200 (29) | 1834000 (22) | 9349000 (23) | 38990000 (31) | 133800000 (17) | 155900000 (17)

15. Secondary Outcome: Part 1: SAD Cohorts: Area Under the Serum Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) for PF-07242813
Description: AUCinf was determined as AUClast + (Clast divided by kel), where Clast = predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel= terminal phase rate constant.
Time Frame: as for outcome 14
Population: The PK parameter set consisted of all randomized participants who received at least 1 dose of study intervention and who have at least 1 of the PK parameters of interest calculated. Here, 'Overall Number of Participants Analyzed' signifies number of participants with evaluable results for this outcome measure. Data was not summarized for PK parameters if less than 3 participants had evaluable data values as pre-specified in the statistical analysis plan.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort)
Number analyzed (Participants) | 0 | 0 | 1 | 6 | 5 | 4 | 5 | 6 | 4
Nanogram*hour/milliliter |  |  | 92700 (NA) — Data for this cohort was not summarized per plan. Individual value for participants was 92700. | 555100 (28) | 1912000 (24) | 9790000 (27) | 46510000 (19) | 153700000 (21) | 173700000 (20)

16. Secondary Outcome: Part 1: SAD Cohorts: Maximum Serum Concentration (Cmax) for PF-07242813
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort)
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4
Nanogram per milliliter | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 38.8 and 67.9. | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 241 and 304. | NA (NA) — Data for this cohort was not summarized per plan. Individual values for participants were 801 and 842. | 3271 (23) | 8397 (48) | 33250 (34) | 110200 (24) | 362000 (11) | 445900 (10)

17. Secondary Outcome: Part 1: SAD Cohorts: Time to Reach Maximum Concentration (Tmax) for PF-07242813
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort)
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 4
Hours | NA [NA to NA] — Data for this cohort was not summarized per plan. Individual values for participants were 2 and 12. | NA [NA to NA] — Data for this cohort was not summarized per plan. Individual values for participants were 0.6 and 2. | NA [NA to NA] — Data for this cohort was not summarized per plan. Individual values for participants were 0.617 and 2. | 2.00 [0.60 to 2.00] | 2.00 [0.60 to 72.00] | 1.61 [1.22 to 12.00] | 2.00 [1.22 to 2.00] | 2.00 [1.22 to 12.00] | 1.22 [1.22 to 1.22]

18. Secondary Outcome: Part 1: SAD Cohorts: Terminal Elimination Half Life (t1/2) for PF-07242813
Description: t1/2 was determined by "Loge(2)/kel", where kel was the terminal phase rate constant calculated by a linear regression of the loglinear -concentration time- curve.
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort)
Number analyzed (Participants) | 0 | 0 | 1 | 6 | 5 | 4 | 5 | 6 | 4
Hours |  |  | NA (NA) — Data for this cohort was not summarized per plan. Individual value for participants was 107. | 138.0 (38.152) | 170.8 (46.300) | 256.0 (65.396) | 434.6 (50.708) | 557.8 (118.48) | 545.5 (80.707)

19. Secondary Outcome: Part 1: MAD Cohorts: Area Under the Serum Concentration Time Profile Over the Dosing Interval (AUCtau) for PF-07242813
Description: Area under the serum concentration time- profile over the dosing interval tau where tau=2 weeks (336 hours).
Time Frame: Day 1,15,29(Pre-dose,2,6,12,24,48,72,96 hours post-dose) Day 15,29(168hours post-dose) Day 29(336hours post-dose) (For all cohorts); Day 1(168hours post-dose for all except 15mg and 50 mg post-dose)
Population: The PK parameter set consisted of all randomized participants who received at least 1 dose of study intervention and who have at least 1 of the PK parameters of interest calculated. Here, 'Number Analyzed' signifies number of participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: Nanogram*hour/milliliter
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram*hour/milliliter
  Day 1 | 296000 (47) | 981600 (46) | 5543000 (23) | 12560000 (36) | 27290000 (24)
  Day 15: number analyzed (Participants) | 6 | 6 | 5 | 5 | 6
  Day 15 | 503400 (39) | 2294000 (37) | 10160000 (4) | 19190000 (20) | 50040000 (28)
  Day 29: number analyzed (Participants) | 6 | 6 | 4 | 4 | 6
  Day 29 | 615300 (39) | 3172000 (32) | 11880000 (14) | 24500000 (13) | 68840000 (27)

20. Secondary Outcome: Part 1: MAD Cohorts: Cmax for PF-07242813
Time Frame: Day 1,15,29(Pre-dose,2,6,12,24,48,72,96 hours post-dose) Day 15,29(168hours post-dose) Day 29(336,672,1008,1344,1680hours post-dose) (For all cohorts); Day 1(168hours post-dose for all except 15mg and 50 mg post-dose)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram per milliliter
  Day 1 | 1087 (43) | 3619 (39) | 21380 (13) | 48550 (36) | 163800 (18)
  Day 15: number analyzed (Participants) | 6 | 6 | 5 | 5 | 6
  Day 15 | 1828 (33) | 8052 (38) | 39470 (19) | 76130 (40) | 266100 (32)
  Day 29: number analyzed (Participants) | 6 | 6 | 4 | 4 | 6
  Day 29 | 1778 (75) | 10470 (33) | 41080 (19) | 83590 (16) | 332900 (20)

21. Secondary Outcome: Part 1: MAD Cohorts: Tmax for PF-07242813
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours
  Day 1 | 96.00 [96.00 to 336.00] | 216.05 [72.00 to 336.00] | 96.00 [72.00 to 146.00] | 72.00 [23.80 to 167.00] | 1.61 [1.22 to 2.00]
  Day 15: number analyzed (Participants) | 6 | 6 | 5 | 5 | 6
  Day 15 | 168.00 [48.00 to 216.00] | 156.00 [144.00 to 336.00] | 96.20 [23.90 to 143.00] | 48.00 [48.00 to 169.00] | 2.00 [1.22 to 2.00]
  Day 29: number analyzed (Participants) | 6 | 6 | 4 | 4 | 6
  Day 29 | 168.50 [48.00 to 171.00] | 157.50 [146.00 to 312.00] | 135.00 [48.00 to 170.00] | 72.60 [23.80 to 148.00] | 4.00 [2.00 to 23.80]

22. Secondary Outcome: Part 1: MAD Cohorts: Terminal Elimination Half Life (t1/2) for PF-07242813
Description: t1/2 was determined by "Loge(2) per kel", where kel was the terminal phase rate constant calculated by a linear regression of the log/linear -concentration time- curve.
Time Frame: as for outcome 20
Population: The PK parameter set consisted of all randomized participants who received at least 1 dose of study intervention and who have at least 1 of the PK parameters of interest calculated. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD
Number analyzed (Participants) | 2 | 6 | 4 | 4 | 4
Hours
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 29 | 111 (190) | 210.5 (82.674) | 352.8 (99.704) | 475.5 (140.58) | 474.0 (98.346)

23. Secondary Outcome: Part 2: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 6
Description: EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Time Frame: Baseline, Week 6
Population: Modified Intention to Treat (mITT) population consisted of all randomized participants assigned to study intervention and who applied at least 1 dose of study intervention. One participant was randomized twice under different participant ID (PID) at two different sites. The participant was included in the efficacy analyses under the first PID. The participant enrolled under the second PID was included in mITT per mITT definition, but was excluded from efficacy analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
Number analyzed (Participants) | 15 | 9
Percent change | -38.2 [-54.2 to -22.2] | -43.8 [-65.3 to -22.3]
Statistical Analysis 1: Comparison: Part 2: 1000 mg IV AD vs Part 2: Placebo IV AD; Test type: Other; p = 0.6343, ANCOVA; Least Square Mean Difference = 5.6, 90% CI 2-sided [-21.4 to 32.6]

ADVERSE EVENTS:
Time Frame: For SAD (From start of study treatment on Day 1 to Day 71), for MAD (From start of study treatment on Day 1 to Day 99), and for AD (From start of study treatment on Day 1 to Week 16).
Description: An AE term may be reported as both a serious and non-serious AE but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Part 1: 0.3 mg IV SAD | Part 1: 1mg IV SAD | Part 1: 3 mg IV SAD | Part 1: 10 mg IV SAD | Part 1: 30 mg IV SAD | Part 1: 100 mg IV SAD | Part 1: 300 mg IV SAD | Part 1: 1000 mg IV SAD | Part 1: 1000 mg IV SAD (Japanese Cohort) | Part 1: 15 mg SC Q2W MAD | Part 1: 50 mg SC Q2W MAD | Part 1: 150 mg SC Q2W MAD | Part 1: 300 mg SC Q2W MAD | Part 1: 500 mg IV Q2W MAD | Part 1: Placebo SAD | Part 1: Placebo SC MAD | Part 1: Placebo IV MAD | Part 2: 1000 mg IV AD | Part 2: Placebo IV AD
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/17 | 0/8 | 0/2 | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 1/17 | 0/8 | 0/2 | 0/16 | 1/9
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/4 | 0/6 | 0/6 | 0/6 | 0/6 | 2/6 | 0/17 | 0/8 | 0/2 | 1/16 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 0.3 mg IV SAD (N=2) | Part 1: 1mg IV SAD (N=2) | Part 1: 3 mg IV SAD (N=2) | Part 1: 10 mg IV SAD (N=6) | Part 1: 30 mg IV SAD (N=6) | Part 1: 100 mg IV SAD (N=6) | Part 1: 300 mg IV SAD (N=6) | Part 1: 1000 mg IV SAD (N=6) | Part 1: 1000 mg IV SAD (Japanese Cohort) (N=4) | Part 1: 15 mg SC Q2W MAD (N=6) | Part 1: 50 mg SC Q2W MAD (N=6) | Part 1: 150 mg SC Q2W MAD (N=6) | Part 1: 300 mg SC Q2W MAD (N=6) | Part 1: 500 mg IV Q2W MAD (N=6) | Part 1: Placebo SAD (N=17) | Part 1: Placebo SC MAD (N=8) | Part 1: Placebo IV MAD (N=2) | Part 2: 1000 mg IV AD (N=16) | Part 2: Placebo IV AD (N=9)
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 0.3 mg IV SAD (N=2) | Part 1: 1mg IV SAD (N=2) | Part 1: 3 mg IV SAD (N=2) | Part 1: 10 mg IV SAD (N=6) | Part 1: 30 mg IV SAD (N=6) | Part 1: 100 mg IV SAD (N=6) | Part 1: 300 mg IV SAD (N=6) | Part 1: 1000 mg IV SAD (N=6) | Part 1: 1000 mg IV SAD (Japanese Cohort) (N=4) | Part 1: 15 mg SC Q2W MAD (N=6) | Part 1: 50 mg SC Q2W MAD (N=6) | Part 1: 150 mg SC Q2W MAD (N=6) | Part 1: 300 mg SC Q2W MAD (N=6) | Part 1: 500 mg IV Q2W MAD (N=6) | Part 1: Placebo SAD (N=17) | Part 1: Placebo SC MAD (N=8) | Part 1: Placebo IV MAD (N=2) | Part 2: 1000 mg IV AD (N=16) | Part 2: Placebo IV AD (N=9)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04668066/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT04668066/SAP_001.pdf